CLINICAL TRIAL: NCT00519948
Title: Comfort and Cleaning Evaluation of Multipurpose Solutions in Contact Lens Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Dr. Chu, Eyeworks Group
Model: Crossover | Masking: None
Other Study IDs: 5320
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Patient Comfort; Lens Cleanliness

INTERVENTIONS:
Drug: new MPS, opti-free express no rub MPS

SUMMARY:
To compare patient comfort and overall lens cleanliness with consecutive use of two multipurpose lens solutions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 yrs or older
2. Males or females
3. Any race or ethnic background
4. CL patients using Opti-Free Express no-rub MPS currently
5. Patients using Focus night and day Lenses

Exclusion Criteria:

1. Corneal refractive surgery within 6 months of this study.
2. Corneal ectasia.
3. Current use of Restasis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Chu, OD, Principal Investigator — Eyeworks Group
Locations (1):
- Eyeworks Group, Fort Worth, Texas, United States